CLINICAL TRIAL: NCT07037433
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Impact of Maridebart Cafraglutide on Cardiovascular Outcomes in Participants With Atherosclerotic Cardiovascular Disease and Overweight or Obesity
Brief Title: Evaluating the Impact of Maridebart Cafraglutide on Cardiovascular Outcomes in Participants With Atherosclerotic Cardiovascular Disease and Overweight or Obesity
Acronym: MARITIME-CV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20220196
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atherosclerotic Cardiovascular Disease; Overweight; Obesity
Keywords: Atherosclerotic Cardiovascular Disease; Overweight; Obesity; Maridebart cafraglutide; AMG 133; MariTide
MeSH Terms: conditions — Atherosclerosis; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maridebart Cafraglutide (Experimental): Participants will receive maridebart cafraglutide subcutaneously (SC).
  Interventions: Drug: Maridebart Cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to demonstrate that maridebart cafraglutide is superior to placebo when given as an adjunct to standard of care with respect to reducing cardiovascular (CV) morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 45 years at screening.
* BMI of ≥ 27 kg/m2 at screening.
* History of Atherosclerotic Cardiovascular Disease (ASCVD) as evidenced by at least one of the following:

  * Prior MI.
  * Prior ischemic stroke (may include ischemic stroke with hemorrhagic transformation).
  * Symptomatic peripheral arterial disease (PAD), as evidenced by intermittent claudication with ankle-brachial index (ABI) < 0.9 (at rest), or peripheral arterial revascularization procedure, or amputation due to atherosclerotic disease.

Exclusion Criteria

* History of any of the following within 60 days before screening: MI, hospitalization for unstable angina, coronary artery revascularization, coronary artery bypass graft surgery or other major cardiovascular surgery, stroke, or transient ischemic attack (TIA).
* New York Heart Association (NYHA) class IV HF at screening or hospitalization for HF within 60 days before screening.
* Type 1 DM, or any type of diabetes with the exception of T2DM or history of gestational diabetes.
* For participants with a prior diagnosis of T2DM at screening:

  * HbA1c > 10.0% (86 mmol/mol) at screening.
  * History of diabetic ketoacidosis or hyperosmolar state/coma within 12 months before screening.
  * One or more episodes of severe hypoglycemia within 6 months before screening and/or history of hypoglycemia unawareness.
  * History of proliferative diabetic retinopathy, diabetic maculopathy, or severe non-proliferative diabetic retinopathy.
* Use of any glucagon-like peptide-1 receptor agonist (GLP-1 RA), glucose-dependent insulinotropic polypeptide (GIP) agonists or antagonists, or amylin analogs within 90 days before randomization or planned use during the conduct of the study.
* History of chronic pancreatitis or history of acute pancreatitis in the 180 days before screening.
* Family (first-degree relative[s]), or personal history of medullary thyroid carcinoma (MTC), or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* Calcitonin ≥ 50 ng/L (pg/mL) at screening.
* Acute or chronic hepatitis; signs and symptoms of any liver disease other than metabolic dysfunction-associated steatotic liver disease, or alanine aminotransferase (ALT) > 3.0 x the upper limit of normal (ULN), or total bilirubin (TBL) > 1.8 x ULN (for participants with a known diagnosis of Gilbert syndrome, direct bilirubin should be used instead of TBL).
* History of malignancy within the last 5 years before screening (except for the following treated with curative intent: non-melanoma skin cancer, breast ductal carcinoma in situ, cervical carcinoma in situ, or prostate cancer in situ).
* Participants of childbearing potential planning to become pregnant while on study or unwilling to use protocol-specified methods of contraception during treatment.

Ages: 45 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12800 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-09-29 (Estimated)

PRIMARY OUTCOMES:
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death, Myocardial Infarction (MI), or Ischemic Stroke (3-point Major Adverse Cardiac Events [3-P MACE]) | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of: All-cause Death, MI, Ischemic Stroke, Coronary Revascularization, or Heart Failure (HF) Event (5-point MACE) | Up to approximately 35 months

SECONDARY OUTCOMES:
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death, MI, Ischemic Stroke, or HF Event | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death, MI, Ischemic Stroke or Coronary Revascularization | Up to approximately 35 months
Time to First MI | Up to approximately 35 months
Time to First Ischemic Stroke | Up to approximately 35 months
Time to CV Death | Up to approximately 35 months
Time to All-cause Death | Up to approximately 35 months
Time to First Coronary Revascularization | Up to approximately 35 months
Time to First HF Event | Up to approximately 35 months
Time to First HF Event or CV Death | Up to approximately 35 months
Time to First Unstable Angina Requiring Hospitalization | Up to approximately 35 months
Time to First Occurrence of MI or CV Death | Up to approximately 35 months
Time to First Occurrence of MI, Ischemic Stroke or All-cause Death | Up to approximately 35 months
Total Major Ischemic Events (Time to First and Recurrent MI or Ischemic Stroke) | Up to approximately 35 months
Total All-cause Hospitalizations (Time to First and Recurrent Event) | Up to approximately 35 months
Time to Onset of Type 2 Diabetes Mellitus (T2DM) in Participants with Prediabetes at Baseline | Up to approximately 35 months
Time to Onset of T2DM in Participants without T2DM at Baseline | Up to approximately 35 months
Change from Baseline in Systolic Blood Pressure (SBP) at Week 72 | Baseline and Week 72
Change from Baseline in Diastolic Blood Pressure (DBP) at Week 72 | Baseline and Week 72
Change from Baseline in Body Mass Index (BMI) at Week 72 | Baseline and Week 72
Change from Baseline in Waist Circumference at Week 72 | Baseline and Week 72
Change from Baseline in Urine Albumin-to-creatinine Ratio (uACR) at Week 72 | Baseline and Week 72
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 72 | Baseline and Week 72
Change from Baseline in Fasting Plasma Glucose at Week 72 | Baseline and Week 72
Percent Change from Baseline in High-sensitivity C-reactive protein (hs-CRP) at Week 72 | Baseline and Week 72
Percent Change from Baseline in Body Weight at Week 72 | Baseline and Week 72
Percent Change from Baseline in Total Cholesterol at Week 72 | Baseline and Week 72
Percent Change from Baseline in High-density Lipoprotein Cholesterol (HDL-C) at Week 72 | Baseline and Week 72
Percent Change from Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Week 72 | Baseline and Week 72
Percent Change from Baseline in Triglycerides (TG) at Week 72 | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 6.5% (48 mmol/mol) in Participants with T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 6.0% (42 mmol/mol) in Participants with T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 5.7% (39 mmol/mol) in Participants with T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 6.5% (48 mmol/mol) in Participants Without T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 6.0% (42 mmol/mol) in Participants Without T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 5.7% (39 mmol/mol) in Participants Without T2DM at Baseline | Baseline and Week 72
Number of Participants at Week 72 with HbA1c < 5.7% (39 mmol/mol) in Participants with HbA1c ≥ 5.7% and < 6.5% at Baseline | Baseline and Week 72
Change from Baseline in Short Form 36 Health Survey Acute Version 2 (SF-36 v2) Physical Function Domain Score at Week 48 | Baseline and Week 48
Time to First Event of a Composite Nephropathy Endpoint | Up to approximately 35 months
  Composite endpoint consists of onset of persistent macroalbuminuria, persistent ≥ 40% reduction in estimated glomerular filtration rate (eGFR), onset of persistent eGFR < 15 mL/min/1.73 m2, initiation of chronic renal replacement therapy (dialysis or transplantation), CV or renal death.
Change in eGFR (total slope) for the period from baseline to the final follow up visit | Baseline up to approximately 35 months
Change in eGFR (chronic slope) for the period from 4 months to the final follow-up visit | From 4 months up to approximately 35 months
Time to First Occurrence of a Major Adverse Limb Event (MALE) Defined as Acute Limb Ischemia, Urgent Peripheral Revascularization, Major Amputation Due to a Vascular Etiology or Chronic Limb-threatening Ischemia Requiring Revascularization | Up to approximately 35 months
Total Arterial (Coronary, Cerebrovascular, and Peripheral) Revascularization Procedures (Time to First and Recurrent Event) | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death, MI, Ischemic Stroke, MALE, or Arterial Revascularization | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of: CV Death, MI, Ischemic Stroke, or Acute Limb Ischemia | Up to approximately 35 months
Time to First Occurrence of a Composite Endpoint Consisting of CV Death, MI, Ischemic Stroke, Acute Limb Ischemia, or Urgent Arterial Revascularization Procedure (Coronary, Cerebrovascular or Peripheral) | Up to approximately 35 months
Number of Participants with Treatment-emergent Adverse Events | Up to approximately 35 months
Number of Participants with Serious Adverse Events | Up to approximately 35 months
Plasma Concentration of Maridebart Cafraglutide at Week 72 | Week 72

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (712):
- United States (134):
  - Alliance For Multispecialty Research - Daphne, Daphne, Alabama
  - Eastern Shore Research Institute, Fairhope, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Mobile Heart Specialists PC, Mobile, Alabama
  - Syed Research Consultants LLC, Sheffield, Alabama
  - Synexus Clinical Research US, Inc., Phoenix, Arizona
  - Medical Advancement Centers of Arizona, Phoenix, Arizona
  - Valley Clinical Trials, LLC dba Flourish Research, Covina, California
  - Velocity Clinical Research- Huntington Park, Huntington Park, California
  - Velocity Clinical Research- Los Angeles, La Mesa, California
  - Orange County Research Center, Lake Forest, California
  - Biopharma Informatic - The Cardiovascular Center, Redding, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Walnut Creek, California
  - Focus Clinical Research, West Hills, California
  - Family Practice Associates, Wilmington, Delaware
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Velocity Clinical Research - New Smyrna Beach, Edgewater, Florida
  - Alliance for Multispecialty Research - Fort Myers, Fort Myers, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Elite Cardiac Research Center LLC, Hialeah, Florida
  - Elite Clinical Research, Hialeah, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Clinical Research of Central Florida, Lakeland, Florida
  - South Florida Clinical Research, Margate, Florida
  - Finlay Medical Research, Miami, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - San Marcus Research Clinic Inc, Miami Lakes, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Saint Johns Center for Clinical Research, Saint Augustine, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - East Coast Institute for Research LLC at Canton Georgia, Canton, Georgia
  - The Jones Center Clinical Research, Macon, Georgia
  - Velocity Clinical Research - Savannah, Savannah, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Eagle Clinical Research, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Alliance For Multispecialty Research - Oak Brook, Oak Brook, Illinois
  - Prarie Education and Research, Springfield, Illinois
  - Cardiovascular Research of Northwest Indiana LLC, Munster, Indiana
  - Velocity Clinical Research - Valparaiso, Valparaiso, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Cotton-ONeil Diabetes and Endocrinology Center, Topeka, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Cardiovascular Associates Research, LLC, Covington, Louisiana
  - Tandem Clinical Research - Marrero, Marrero, Louisiana
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Velocity Clinical Research - Rockville, Rockville, Maryland
  - Btc of New Bedford, New Bedford, Massachusetts
  - Fairview Health Services M Health Fairview St Johns Hospital, Maplewood, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Saint Louis Heart and Vascular PC, St Louis, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Primary Clinical Research, Papillion, Nebraska
  - Alliance Clinical Research, Las Vegas, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - CardioMetabolic Collaborative Clinic, Somerset, New Jersey
  - Velocity Clinical Research - Binghamton, Binghamton, New York
  - Hudson Valley Cardiovascular Practice PC, Poughkeepsie, New York
  - Rochester Clinical Research, Rochester, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Southgate Medical Group, West Seneca, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Velocity Clinical Research - Durham, Durham, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Burke Primary Care Family Practice, Morganton, North Carolina
  - Accellacare of Raleigh, Raleigh, North Carolina
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - Brookview Hills Research Associates Llc, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Aultman Hospital, Cardiovascular Consultants, Inc, Canton, Ohio
  - Velocity Clinical Research - Auburn, Cincinnati, Ohio
  - Endocrinology Associates Inc, Columbus, Ohio
  - Nexgen Research, Lima, Ohio
  - Alliance for Multispecialty Research - Norman, Norman, Oklahoma
  - Heritage Valley Multispecialty Group Inc, Beaver, Pennsylvania
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - Abington Medical Specialists, Horsham, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Accellacare Charleston, Mt. Pleasant, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Stern Cardiovascular Foundation Inc, Germantown, Tennessee
  - Accellacare of Knoxville, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville North Knoxville Medical Center, Powell, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - PharmaTex Research, LLC, Amarillo, Texas
  - Austin Heart, Austin, Texas
  - Velocity Clinical Research - Austin, Austin, Texas
  - Thyroid Endocrinology and Diabetes, Dallas, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Cedar Health Research, LLC, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - David Turbay, MD, El Paso, Texas
  - Academy of Diabetes Thyroid and Endocrine, El Paso, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Cardiovascular Specialists of Willowbrook, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Research Physicians Network, LLC, Houston, Texas
  - Vital Heart and Vein, Humble, Texas
  - Tcr Institute Llc, Kingwood, Texas
  - Helium Research Group, Lake Jackson, Texas
  - Epic Clinical Research, Lewisville, Texas
  - Biopharma Informatic-McAllen, McAllen, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - North Hills Medical Research, North Richland Hills, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Consano Clinical Research - Shavano Park, Shavano Park, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - Boeson Research, Provo, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Inova Cardiology - Fairfax, Fairfax, Virginia
  - Velocity Clinical Research - Spokane, Spokane, Washington
  - Vaught Neurological Services, Crab Orchard, West Virginia
  - Aspirus Cardiovascular Associates, Wausau, Wisconsin
- Argentina (25):
  - Centro Medico Viamonte, CABA, Buenos Aires
  - Imoba Investigaciones medicas, CABA, Buenos Aires
  - Conexa Investigacion Clinica SA, CABA, Buenos Aires
  - Stat Research, CABA, Buenos Aires
  - Cedic - Centro de Investigacion Clinica, CABA, Buenos Aires
  - Cemedic Centro de Especialidades Medicas, CABA, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, CABA, Buenos Aires
  - Consultorios Medicos Dr Besada, CABA, Buenos Aires
  - Fundacion Respirar - Consultorios Medicos Dr Doreski, CABA, Buenos Aires
  - Glenny Corp SA, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Ciprec - Centro de Investigacion y Prevencion Cardiovascular, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas de San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Go Centro Medico San Nicolas, Zárate, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - Centro Diabetologico Dr Waitman, Córdoba, Córdoba Province
  - Clinica Privada del Prado, Córdoba, Córdoba Province
  - Instituto Medico Rio Cuarto SA, Río Cuarto, Córdoba Province
  - mit - Medicina Investigacion y Tratamiento, Santa Rosa, La Pampa Province
  - CIPADi, Godoy Cruz, Mendoza Province
  - Instituto Medico Catamarca Imec, Rosario, Santa Fe Province
  - Centro Medico de Nutricion y Diabetes, CABA
  - INECO Neurociencias Oronio, Rosario
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Australia (16):
  - Novatrials, Charlestown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Momentum Clinical Research - Darlinghurst, Sydney, New South Wales
  - Advara HeartCare Wesley, Auchenflower, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Dr Heart Pty Ltd, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Advara HeartCare Leabrook, Leabrook, South Australia
  - Victorian Heart Hospital, Clayton, Victoria
  - Barwon Health Geelong Hospital, Geelong, Victoria
  - Austin Health, Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Advara HeartCare Mulgrave, Mulgrave, Victoria
  - Advara HeartCare Joondalup, Joondalup, Western Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Medizinische Universitaet Graz, Graz
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Krankenhaus der Barmherzigen Brueder Linz, Linz
  - Klinik Landstrasse, Vienna
  - Zentrum fuer klinische Studien - Dr Hanusch GmbH, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (12):
  - Azorg Campus Aalst - Moorselbaan, Aalst
  - Imelda Ziekenhuis vzw, Bonheiden
  - Algemeen Ziekenhuis Sint-Jan Brugge, Bruges
  - Cliniques universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - Algemeen Ziekenhuis Sint Lucas, Ghent
  - Centres Hospitaliers Universitaires - Helora - Hopital de La Louviere - Site Jolimont, La Louvière
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - AZ Oostende - Damiaan, Ostend
  - Universite Catholique de Louvain Cliniques Universitaires de Mont-Godinne, Yvoir
- Brazil (35):
  - Centro de Pesquisas em Diabetes e Doencas Endocrino Metabolicas, Fortaleza, Ceará
  - Centro do Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Inovace Pesquisa Clinica, Salvador, Estado de Bahia
  - Instituto de Ensino e Pesquisa do Hospital do Coracao do Brasil, Brasília, Federal District
  - Assoc Amparo Saude Ensin e Pesquisa, Brasília, Federal District
  - NS Clinica De Endocrinologia E Diabetes - Cendi, Goiânia, Goiás
  - Hospital das Clinicas da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Universitario Maria Aparecida Pedrossian, Campo Grande, Mato Grosso do Sul
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Ccih - Consultoria em Controle de Infecção Hospitalar, Belo Horizonte, Minas Gerais
  - Cardresearch Cardiologia Assistencial de Pesquisa, Belo Horizonte, Minas Gerais
  - Eurolatino Pesquisas Medicas, Uberlândia, Minas Gerais
  - Quanta Diagnostico por Imagem, Curitiba, Paraná
  - Hospital Universitário João de Barros Barreto, Belém, Pará
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - Instituto Atena de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - jmf Clinica do Coracao ltda, Aracaju, Sergipe
  - Loema Instituto de Pesquisa Clinica e Consultores Ltda - Clinica Loema, Campinas, São Paulo
  - Instituto de Pesquisa Clinica de Campinas - Ipecc, Campinas, São Paulo
  - Instituto do Coracao de Marilia, Marília, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - Cemec Centro Multidisciplinar Estudos Clinicos, São Bernardo do Campo, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Ispem - Instituto Sao Jose dos Campos em Pesquisas Medicas, São José dos Campos, São Paulo
  - Centro de Pesquisas Clinicas Cpclin, São Paulo, São Paulo
  - Instituto de Molestias Cardiovasculares de Tatui, Tatuí, São Paulo
  - IBPClin Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Ruschel Medicina e Pesquisa Clinica, Rio de Janeiro
  - Br Trials - Ensaios Clínicos e Consultoria, São Paulo
  - CPQuali Pesquisa Clinica Ltda, São Paulo
  - Centro Paulista de Investigacao Clinica Cepic, São Paulo
  - Instituto do Coracao do Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Bulgaria (10):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - Medical Center Doctor Staikov EOOD, Burgas
  - Medical Center Medconsult Pleven OOD, Pleven
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - Multiprofile Hospital for Active Treatment Sveta Karidad EAD, Plovdiv
  - National Multiprofile Transport Hospital Tzar Boris III, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Military Medical Academy - Multiprofile Hospital for Active Treatment Sofia, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N I Pirogov EAD, Sofia
  - Medical Center Dr Kalchev OOD, Sofia
- Canada (16):
  - Janek Senaratne Professional Medical Corporation, Edmonton, Alberta
  - Vancouver General Hospital, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Discovery Clinical Services Ltd, Victoria, British Columbia
  - G A Research Associates Limited, Moncton, New Brunswick
  - Centricity Research Brampton, Brampton, Ontario
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - KMH Cardiology Centres Incorporated Hamilton, Stoney Creek, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l Universite de Montreal, Montreal, Quebec
  - Research Institute of McGill University Health Center - Glen Site, Montreal, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - Centre intégré de santé et service sociaux de Lanaudière, Saint-Charles-Borromée, Quebec
- China (38):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou Central Peoples Hospital, Huizhou, Guangdong
  - The First Peoples Hospital of Yulin, Yulin, Guangxi
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science And Technology, Luoyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi Peoples Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - China Japan Union Hospital of Jilin University, Changchun, Jilin
  - Shaanxi Provincial Peoples Hospital, Xi'an, Shaanxi
  - Xi'an Daxing Hospital, Xi'an, Shaanxi
  - Jinan Central Hospital, Jinan, Shandong
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tenth Peoples Hospital, Shanghai, Shanghai Municipality
  - The Fifth Peoples Hospital of Shanghai, Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi An Jiao Tong University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Chengdu Fifth Peoples Hospital, Chengdu, Sichuan
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Sichuan
  - Tianjin Peoples Hospital, Tianjin, Tianjin Municipality
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
- Czechia (40):
  - Innera sro, Benešov
  - Medicentrum Beroun as, Beroun
  - MUDr Libor Nechvatal sro, Brno
  - Centrum pro zdravi sro, Brno
  - MUDr Karel Kamenik sro, Brno
  - Kardiologicka ambulance Brno sro, Brno
  - Fakultni nemocnice Brno, Brno
  - Vojenska nemocnice Brno, Brno
  - Amkardia sro, Brno
  - CorMedico sro, Bruntál
  - Kardio Chlumec sro, Chlumec nad Cidlinou
  - Ordinace pro choroby srdce sro, Chomutov
  - Dika centrum sro, Havirov - Mesto
  - Edumed sro, Hradec Králové
  - Nemocnice Jihlava po, Jihlava
  - Interna a diabetologie MUDr Vodickova sro, Liberec
  - Kardiologie - Liberec sro, Liberec
  - Edumed sro, Náchod
  - Interni a diabetologicka ordinace sro, Náchod
  - PreventaMed sro, Olomouc
  - Ostin sro, Ostrava
  - CCR Ostrava sro, Ostrava
  - MUDr Miroslav Koliba sro, Ostrava
  - Diahelp sro, Pardubice
  - Pratia Pardubice as, Pardubice
  - Kardiologie a Angiologie Praha sro - Komplexni Centrum Vyzkumu, Prevence a Lecby Kardiov Nemoci, Prague
  - Kardiologie a angiologie sro, Prague
  - Avicena - kardiologie, interna sro, Prague
  - Kardiologie Vinohrady sro, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Milan Kvapil sro, Prague
  - Restrial sro, Prague
  - Endokrinologie Cerny Most sro, Prague
  - Kardiologie Cor sro, Praha 10 - Zabehlice
  - MUDr Jarmila Otrubova, Prostějov
  - Kardio Vaclavik sro, Přerov
  - Nemocnice Slany, Slaný
  - MUDrych sro, Svitavy
  - Clinical Trials Service sro, Uherské Hradiště
  - Kardiologie - Usti nad Labem sro, Ústí nad Labem
- Denmark (13):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Esbjerg sygehus Syddansk universitetshospital, Esbjerg
  - Sanos Gandrup, Gandrup
  - Steno Diabetes Center Copenhagen, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Holbaek Sygehus, Holbæk
  - Hvidovre Hospital, Hvidovre
  - Frederiksberg Hospital, København NV
  - Amager Hospital, København S
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Svendborg Sygehus, Svendborg
  - Sanos Vejle, Vejle
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Studycor Oy, Jyväskylä
  - Health Step Finland, Kuopio
  - Oulu University Hospital, Oulu
  - Tays sydankeskus oy, Tampere
- France (16):
  - Centre Hospitalier Regional Universitaire de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Dijon - Hopital Francois Mitterrand, Dijon
  - Centre Hospitalier Universitaire de Grenoble - Hopital Nord Michallon, Grenoble
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hopital le Creusot, Le Creusot
  - Centre Hospitalier Saint Joseph Saint Luc, Lyon
  - Hopital de la Conception, Marseille
  - Centre Hospitalier Universitaire de Nice - Hopital Pasteur, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat Claude Bernard, Paris
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Haut Leveque, Pessac
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Regional Universitaire de Strasbourg - Hopital de Hautepierre, Strasbourg
  - Centre Hospitalier Universitaire de Toulouse - Hopital Rangueil, Toulouse
  - Polyclinique Vauban, Valenciennes
  - Centre Hospitalier Universitaire de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (34):
  - Kardiologische Praxis Dr med Wolfgang Jungmair, Bad Homburg
  - Universitaetsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Charite - Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Diabetespraxis Dr. Hermann Braun, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow, Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil gGmbH, Bochum
  - Universitaetsklinikum Bonn, Bonn
  - Klinikum Lippe, Detmold
  - Diabeteszentrum Dortmund, Dortmund
  - Sankt-Johannes-Hospital, Dortmund
  - Cardiologicum Dresden und Pirna Facharztpraxis für Kardiologie und Angiologie, Dresden
  - Universitaetsklinikum Dresden, Dresden
  - Zentrum fuer Klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - Praxis am Markt Dr. Bernd Becker, Essen
  - Unterfrintroper Hausarztzentrum, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - ClinPhenomics CVC GmbH, Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Cardiologicum Hamburg GbR, Hamburg
  - Diabeteszentrum Hamburg West, Hamburg
  - Braun Ambulantes Herzzentrum Kassel, Kassel
  - Universitaetsklinikum Leipzig, Leipzig
  - AmBeNet GmbH, Leipzig
  - Universitaetsklinikum Schleswig-Holstein - Luebeck, Lübeck
  - Kardiologische Praxis Doktor Jens Taggeselle, Markkleeberg
  - Klinikum rechts der Isar der TUM, München
  - Centrum für Diagnostik und Gesundheit, München
  - Zentrum fuer Diabtes und Gefaesskrankheiten im Franziskus Carré Muenster, Münster
  - Universitaetsklinikum Muenster, Münster
  - Praxis Segner - Dr. Braun - Kirsch, Oberwürzbach
  - Red-Institut GmbH, Oldenburg
  - Kardiologische Gemeinschaftspraxis Papenburg, Papenburg
  - Praxis Reinfeld Mitte Dr Joachim Weimer und Dr Katharina Pfeiffer, Reinfeld (Holstein)
  - Praxis Dr med Ayham Al-Zoebi Facharzt fuer Innere Medizin und Kardiologie, Wermsdorf
- Greece (14):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Athens Naval Hospital, Athens
  - General Hospital for Thoracic Diseases of Athens "Sotiria", Athens
  - General Hospital for Thoracic Diseases of Athens "Sotiria, Athens
  - General Hospital of Athens Ippokrateio, Athens
  - General Hospital of Athens Laiko, Athens
  - Alexandra Hospital, Athens
  - Attikon Hospital, Athens
  - Hygeia Hospital, Athens
  - General Hospital Asklipieio Voulas, Athens
  - University Hospital of Ioannina, Ioannina
  - Ahepa University Hospital, Thessaloniki
  - University General Hospital of Thessaloniki Ahepa, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, The University of Hong Kong, Hong Kong
  - Prince of Wales Hospital, Chinese University of Hong Kong, Shatin, New Territories
- Hungary (30):
  - Lausmed Kft, Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Tagore Medical Center, Balatonfüred
  - Dr Lakatos Ferenc Private Cardiology Practice, Békéscsaba
  - Trial Pharma Kft, Budapest
  - Clinexpert Kft, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - PVN Kutato Kft, Budapest
  - Semmelweis Egyetem Varosmajori Sziv- es Ergyogyaszati Klinika, Budapest
  - Eszak-Pesti Centrum Korhaz - Honvedkorhaz, Budapest
  - Budapesti Uzsoki Utcai Korhaz, Budapest
  - Zugloi Egeszsegugyi Szolgalat, Budapest
  - Strazsahegy Medicina Bt, Budapest
  - Borvo Clinic Kft, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Obudai Egeszsegugyi Centrum Kft, Dunaújváros
  - Gyongyosi Bugat Pal Korhaz, Gyöngyös
  - BKS Research Kft, Hatvan
  - Obudai Egeszsegugyi Centrum Kft, Kaposvár
  - Trial Pharma Kft, Kecskemét
  - Komaromi Selye Janos Korhaz, Komárom
  - Borsod-Abauj-Zemplen Varmegyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - IPR Hungary Kft, Miskolc
  - Borbanya Praxis Egeszsegugyi Kft, Nyíregyháza
  - Dr Nagy Laszlo Kardiologiai maganrendeles es SMO, Orosháza
  - COROMED-SMO Kft, Pécs
  - DaVinci Maganklinika, Pécs
  - KomplexLabor Diagnosztika Kft, Szeged
  - Complex Rendelo Med Zrt, Székesfehérvár
  - Obudai Egeszsegugyi Centrum Kft, Zalaegerszeg
- Italy (12):
  - Azienda Unita Locale Socio Sanitaria Berica 8 Ospedale Cazzavillan, Arzignano
  - Azienda Ospedaliera Sant Anna e San Sebastiano, Caserta
  - Casa della salute Ceccano Ospedale, Ceccano
  - Ospedale Santissima Annunziata, Chieti
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Azienda Sanitaria Locale Abruzzo 1 Avezzano, Sulmona e L'Aquila - Ospedale regionale San Salvatore, L’Aquila
  - IRCCS Ospedale San Raffaele, Milan
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Unita Sanitaria Locale Romagna, Rimini
  - Policlinico Universitario Campus Biomedico, Roma
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (29):
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Sapporo, Hokkaido
  - Nakakinen Clinic, Naka, Ibaraki
  - JA Toride Medical Center, Toride-shi, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Tenyoukai Central Clinic, Kagoshima, Kagoshima-ken
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - KKR Tohoku Kosai Hospital, Sendai, Miyagi
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Oita Red Cross Hospital, Ōita, Oita Prefecture
  - Okayama Rosai Hospital, Okayama, Okayama-ken
  - Saiseikai Senri Hospital, Suita-shi, Osaka
  - Medical corporation Sekishin-kai Saitama Sekishinkai Hospital, Sayama-shi, Saitama
  - Sayama Renal Clinic, Sayama-shi, Saitama
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu, Shizuoka
  - Medical Corporation Kenshinkai Minamino Cardiovascular Hospital, Hachioji-shi, Tokyo
  - Affiliated Central Clinic of Higashiyamato Hospital, Higashiyamato-shi, Tokyo
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - NewHeart Watanabe Institute, Suginami-ku, Tokyo
  - Sanin Rosai Hospital, Yonago-shi, Tottori
  - Tokuyama Central Hospital, Shunan-shi, Yamaguchi
- Netherlands (31):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo
  - EB Medical Research, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amsterdam Universitair Medisch Centrum, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf Gasthuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Ziekenhuis location Dordwijk, Dordrecht
  - Albert Schweitzer Ziekenhuis, Locatie Dordwijk, Dordrecht
  - Catharina Ziekenhuis, Eindhoven
  - Spaarne Gasthuis, locatie Haarlem Zuid, Haarlem
  - Sint Jansdal Ziekenhuis, Harderwijk
  - Elkerliek Ziekenhuis, Helmond
  - Tergooiziekenhuizen, locatie Hilversum, Hilversum
  - Bethesda Diabetes Research Center, Hoogeveen
  - Frisius Medisch Centrum, locatie Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - D and A Research and Genetics, Sneek
  - Haga Ziekenhuis, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Universitair Medisch Centrum Utrecht, Utrecht
  - VieCuri Medisch Centrum, Venlo
- Poland (38):
  - Niepubliczny Zaklad Opieki Zdrowotnej Vita Diabetica Malgorzata Buraczyk, Bialystok
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Bielsko-Biala
  - Centrum Medyczne Kermed - Renata Bijata-Bronisz i Ewa Kowalinska Spolka Jawna, Bydgoszcz
  - Centrum Medyczne Lukamed Spzoo, Chojnice
  - American Heart of Poland Spolka Akcyjna, Chrzanów
  - Etg Lublin Spzoo, Dębica
  - Futuremeds Spolka z ograniczona odpowiedzialnoscia, Gdynia
  - Emc Silesia Spolka z ograniczona odpowiedzialnoscia, Katowice
  - Salvia-Lekston i Madej Spolka Jawna, Katowice
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Kędzierzyn-Koźle
  - Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne Diab-Endo-Met Sp zoo, Krakow
  - Unicardia And Unimedica And Uniestetica, Krakow
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Krakow
  - Beata Miklaszewicz i Dariusz Dabrowski Cardiamed Spolka Jawna, Legnica
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Lodz
  - Clinical Best Solutions Sp zoo Spolka Komandytowa Gabinet Lekarski, Lublin
  - Ekamed Spolka z Ograniczona Odpowiedzialnoscia, Lublin
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Olsztyn
  - Uniwersytecki Szpital Kliniczny w Opolu, Opole
  - G and G Medvision Spolka z ograniczona odpowiedzialnoscia, Oświęcim
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Centrum Medyczne Medyk Spolka z Ograniczona Odpowiedzialnoscia Spolka Komandytowa, Rzeszów
  - Nowe Zdrowie-Ck Kieltucki i Wspolnicy Spolka Jawna, Staszów
  - Osrodek Badan Klinicznych Labmed Sp zoo, Szczecin
  - Centrum Szybkiej Diagnostyki Kardiologicznej Kardiomed M Zabowka E Zabowka Spolka cywilna, Tarnów
  - Metabolica Spolka z Ograniczona Odpowiedzialnoscia, Tarnów
  - Praktyka Lekarska Lidia Pawlowicz, Torun
  - Wojewodzki Szpital Zespolony im L Rydygiera w Toruniu, Torun
  - American Heart of Poland Spolka Akcyjna Polsko-Amerykanskie Kliniki Serca, Tychy
  - Futuremeds Spolka z ograniczona odpowiedzialnoscia, Warsaw
  - Clinical Best Solutions Sp zoo Spolka komandytowa, Warsaw
  - Szpital Grochowski imienia Doktora medycyny Rafala Masztaka Spzoo, Warsaw
  - Narodowy Instytut Kardiologii Stefana Kardynala Wyszynskiego Panstwowy Instytut Badawczy, Warsaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SPZOZ we Wroclawiu, Wroclaw
  - Futuremeds spolka z ograniczona odpowiedzialnoscia, Wroclaw
  - Velocity Nova Sp zoo Velocity Zamosc, Zamość
  - Halina Serafin NZOZ Centrum Medyczne "Serafin-Med", Żarów
- Portugal (9):
  - Unidade Local de Saude de Braga, EPE, Braga
  - Unidade Local de Saude de Lisboa Ocidental, EPE - Hospital de Santa Cruz, Carnaxide
  - Unidade Local de Saude de Coimbra, EPE, Coimbra
  - Unidade Local de Saude do Alto Ave, EPE, Guimarães
  - Unidade Local de Saude de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - Unidade Local de Saude de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality
  - Ucardio - Centro Clinico Cardiovascular, Riachos, Torres Novas
  - Unidade Local de Saude de Entre Douro e Vouga, EPE - Hospital de Sao Sebastiao, Santa Maria da Feira
  - Unidade Local de Saude de Gaia-Espinho, EPE, Vila Nova de Gaia
- Research and Cardiovascular, Ponce, Puerto Rico
- Romania (15):
  - Cardioplus Center SRL, Baia Mare
  - cmi Pop Lavinia, Baia Mare
  - Mariodiab Clinic SRL, Brasov
  - Thera Card SRL, Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed, Brasov
  - Geea Medical Easy Diet, Bucharest
  - Centrul pentru Studiul Metabolismului - Hightech Medical Services SRL, Bucharest
  - Institutul National de Diabet si Nutritie si Boli Metabolice N C Paulescu, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Milena Sante, Galati
  - Consultmed SRL, Iași
  - Diabdana SRL, Oradea
  - Clinica Korall, Satu Mare
  - Mediab SRL, Târgu Mureş
  - Cabinet Medical Individual Dr Podoleanu Cristian, Târgu Mureş
- Singapore (6):
  - Sengkang General Hospital, Singapore, Sengkang
  - National University Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
- Slovakia (18):
  - Alian, sro, Bardejov
  - MediTask, sro, Bratislava
  - Novate sro, Bratislava
  - Medispektrum sro, Bratislava
  - Medical group Kosice sro, Košice
  - Cardio D and R, sro Kosice, Košice
  - Kardio 1 sro, Lučenec
  - MediVet, sro, Malacky
  - Nemocnicna as, Malacky
  - Nemocnica s poliklinikou Stefana Kukuru Michalovce, as, Michalovce
  - Oralek, sro, Námestovo
  - InterStom, sro, Nitra
  - Intermedis sro, Prešov
  - Medispol, sro, Prešov
  - Tatratrial sro, Rožňava
  - Medi-Dia sro, Sabinov
  - Interna SK, sro, Svidník
  - Pentes, sro, Žilina
- South Korea (13):
  - Keimyung University Dongsan Medical Center, Daegu
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon-do
- Spain (32):
  - Hospital Vithas Sevilla, Castilleja de la Cuesta, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Complejo Hospitalario de Jaen, Jaén, Andalusia
  - Hospital QuironSalud Malaga, Málaga, Andalusia
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Nuevas Tecnologias en Diabetes y Endocrinologia, Seville, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital Clinic i Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Universitari Sant Joan de Reus, Reus, Catalonia
  - Hospital Universitario de Badajoz, Badajoz, Extremadura
  - Complexo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Complexo Hospitalario Universitario de Ferrol Hospital Universitario Arquitecto Marcide, Ferrol, Galicia
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, Galicia
  - Hospital Alvaro Cunqueiro, Vigo, Galicia
  - Hospital Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de La Ribera, Alzira, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario de Leon, León
  - FutureMeds Madrid, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Sanitas la Zarzuela, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Sweden (7):
  - Falu Lasarett, Falun
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Linkopings Universitetssjukhus, Linköping
  - Clemenstorgets Hjartmottagning, Lund
  - Orebros Universitetssjukhus, Örebro
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Switzerland (5):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Istituto Cardiocentro Ticino, Lugano
  - Universitaetsspital Zuerich, Zurich
- Taiwan (7):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital of Chang Gung Medical Foundation, Taoyuan District
- Turkey (Türkiye) (15):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Afyonkarahisar Saglik Bilimleri Universitesi Hastanesi, Afyonkarahisar
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Bursa Yuksek Ihtisas Egitim ve Arastirma Hastanesi, Bursa
  - Pamukkale Universitesi Tip Fakultesi Hastanesi, Denizli
  - Koc Universitesi Hastanesi, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bagcilar Medipol Mega Universite Hastanesi, Istanbul
  - Sultangazi Haseki Egitim ve Arastirma Hastanesi, Istanbul
  - Goztepe Prof Dr Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi Hastanesi, Kocaeli
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Samsun
- United Kingdom (26):
  - Heartlands Hospital, Birmingham
  - Waterloo Medical Centre, Blackpool
  - Southmead Hospital, Bristol
  - West Walk Surgery, Bristol
  - Addenbrookes Hospital, Cambridge
  - Countess of Chester Hospital, Chester
  - University Hospital Coventry, Coventry
  - Ninewells Hospital and Medical School, Dundee
  - Staploe Medical Centre, Ely
  - Royal Devon and Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Wycombe Hospital, High Wycombe
  - Hull Royal Infirmary, Hull
  - Glenfield Hospital, Leicester
  - Queen Mary University of London, London
  - Chelsea and Westminster Hospital, London
  - St Georges Hospital, London
  - Northenden Group Practice, Manchester
  - Newcastle NIHR Commercial Research Delivery Centre, Newcastle
  - University Hospital Llandough, Penarth
  - Lister Hospital, Stevenage
  - Morriston Hospital, Swansea
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay
  - Bradford on Avon and Melksham Health Partnership, Wiltshire
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com